CLINICAL TRIAL: NCT02868957
Title: Standardization of Evaluation Protocol for the Performance Comparison of Digital Intra-oral Scanners
Brief Title: Repetition Improves Precision and Trueness of Digital Intraoral Scans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Gwanak Dental Hospital (Other)
Responsible Party: Principal Investigator, Ji-Man Park, Clinical Associate Professor, Seoul National University Gwanak Dental Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ECT14-02A-27; 10053907 (Other Grant/Funding Number: Ministry of Trade, Industry and Energy); NRF-2013R1A1A1076022 (Other Grant/Funding Number: Ministry of Science, ICT & Future Planning)
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Tooth Diseases
Keywords: CAD; Digital imaging; Prosthetic Dentistry
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Impression data from reference scanner (Active Comparator): desktop scanner was used as a reference scanner. According to the data of the manufacturer, the accuracy is less than 20 µm and the scan points more than 100,000.
  Interventions: Device: iTero; Device: Trios
- Trios (Experimental): Trios is a scanner with real time rendering type adopting the confocal principle, and scans the object while showing the scanned area on a screen.
  Interventions: Assigned intervention to participants in this clinical study was in the form of repetitive learning of Trios intra-oral scanner.
  Interventions: Other: impression data from reference scanner; Device: Trios
- iTero (Experimental): iTero captures teeth and periodontal soft tissue using a red laser beam and parallel confocal imaging technology. This system with a focal depth of 300 can capture up to 100,000 of laser points, and each of such laser points is separated at a 50 mm gap.
  Interventions: Assigned intervention to participants in this clinical study was in the form of repetitive learning of iTero intra-oral scanner.
  Interventions: Other: impression data from reference scanner; Device: iTero

INTERVENTIONS:
Other: impression data from reference scanner — To create a reference images for the assessment of the trueness, the impressions of the upper and lower arch of the oral cavities of four patients were taken using a polyether impression material (3M ESPE Soft Monophase; Minnesota Mining and Manufacturing Co.), and the intaglio scanning was performed on the impression body using a desktop scanner. Scanned images were transformed to the Standard Tessellation Language (STL) file format, and used as reference images.
  Arms: Trios; iTero
Device: iTero — The participants visited the dental clinic and performed scanning for 4 days. In order to investigate the difference in the precision and trueness of iTero intraoral scanners, the participants scanned the dental arch of a single patient 10 times using an assigned digital intraoral scanner.
  Arms: Impression data from reference scanner; iTero
Device: Trios — The participants visited the dental clinic and performed scanning for 4 days. In order to investigate the difference in the precision and trueness of Trios intraoral scanners, the participants scanned the dental arch of a single patient 10 times using an assigned digital intraoral scanner. .
  Arms: Impression data from reference scanner; Trios

SUMMARY:
The objectives of this study were to compare the precision of two digital intraoral scanners from a series of repeat scan images, and to investigate the effect of the learning curve on changes in trueness when scanning the full arch of the oral cavity in actual patients.

DETAILED DESCRIPTION:
Study Participants: This study was approved by the institutional review board of Ehwa Womans University Medical Center Mokdong Hospital, and dental hygienists who were suitable for the purpose of the study were selected (ECT14-02A-27). Participants were assigned one of four patients, and subsequently scanned the oral cavity of a single patient 10 times repeatedly over 4 days.

Study Design: The participants visited the dental clinic and performed scanning for 4 days. In order to investigate the difference in the precision and trueness of two types of intraoral scanners, the participants scanned the dental arch of a single patient 10 times using an assigned digital intraoral scanner. On the first day, either of the two types of scanners (iTero and Trios), and a patient were assigned. Then, the participants were trained in theory and practices of the assigned scanner, and subsequently, using it, scanned the dental arch of the assigned patient twice. On the second and third days, the dental arch of the same patient was scanned 3 times respectively, and on the fourth day, the experiment was finished after scanning the same patient twice.

Statistical Analyses: Collected data were analyzed using the SPSS Ver. 20.0 statistical package. For the determination of differences in the deviations according to the scanner, the independent two-sample t-test was conducted to examine the significance of the precision data. For comparisons of trueness according to repeated learning, the repeated measure ANOVA was used to test for differences between the scanners, clinical experience of the participants, and the scanning region within the same scanner group. The significance of time-dependent changes, and the interaction between the scanner group and time variables, were examined by within-subject tests. Differences between the scanner groups were examined by between-subject tests. The significance of the 10 consecutive scans and four visits within the scanner group, and the difference between the scanner groups at each time point, were examined by the post-hoc test, which was performed using the Bonferroni method as a multiple comparison (α= 0.05).

ELIGIBILITY:
Inclusion Criteria:

* The selection criteria for the participants were as follows: they had the clinical experiences between 3 - 11 years, understood the purpose of the study well, gave their consent, and were able to carry out a 4-day learning course. Those who were inadequate to carry out the study mentally or physically.

Exclusion Criteria:

* Applicant who was considered inappropriate .for this study by the principal investigator was excluded from the selection

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Precision and trueness of intraoral scanners after repeated scanning practice assessed by Geomagic Verify Ver.20152.0 | One year
  Assessment was done by registering pairs of scan images and calculating deviation by computer calculation in micrometers.

SECONDARY OUTCOMES:
Scan time required for full arch image acquisition in seconds | up to one year
  Scan time was measured until the scanned image was satisfactory with reference to the standard quality by one inspector.

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Man Park, PhD, Principal Investigator — Seoul National University Gwanak Dental Hosipital
Locations (1):
- Seoul National University Gwanak Dental Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The three dimensional data in .stl format and the time required for the full arch intra-oral scan of the patient will be provided. These data can be provided after the approval of uploaded documents for our clinical trial. The data can be provided via shared files to the individuals who want IPD in this study.

REFERENCES:
- [Background] Lee SJ, Gallucci GO. Digital vs. conventional implant impressions: efficiency outcomes. Clin Oral Implants Res. 2013 Jan;24(1):111-5. doi: 10.1111/j.1600-0501.2012.02430.x. Epub 2012 Feb 22. PMID 22353208
- [Background] Ender A, Mehl A. Influence of scanning strategies on the accuracy of digital intraoral scanning systems. Int J Comput Dent. 2013;16(1):11-21. English, German. PMID 23641661
- [Background] Feldman LS, Cao J, Andalib A, Fraser S, Fried GM. A method to characterize the learning curve for performance of a fundamental laparoscopic simulator task: defining "learning plateau" and "learning rate". Surgery. 2009 Aug;146(2):381-6. doi: 10.1016/j.surg.2009.02.021. Epub 2009 Jun 25. PMID 19628099
- [Background] Yuzbasioglu E, Kurt H, Turunc R, Bilir H. Comparison of digital and conventional impression techniques: evaluation of patients' perception, treatment comfort, effectiveness and clinical outcomes. BMC Oral Health. 2014 Jan 30;14:10. doi: 10.1186/1472-6831-14-10. PMID 24479892
- [Background] Patzelt SB, Lamprinos C, Stampf S, Att W. The time efficiency of intraoral scanners: an in vitro comparative study. J Am Dent Assoc. 2014 Jun;145(6):542-51. doi: 10.14219/jada.2014.23. PMID 24878708